CLINICAL TRIAL: NCT03444857
Title: Effect of Continuous Positive Airway Pressure (CPAP) for Obstructive Sleep Apnea (OSA) on Myocardial Salvage After Primary Percutaneous Coronary Intervention for Acute ST-Segment Elevation Myocardial Infarction: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: CPAP for OSA on Myocardial Salvage After pPCI for STEMI Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Director, Emergency & Critical Care Center, Professor of Medicine, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018006
Record Dates: First submitted 2018-02-20; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Obstructive Sleep Apnea; ST Elevation Myocardial Infarction
Keywords: Continuous Positive Airway Pressure; Myocardial Salvage; Obstructive Sleep Apnea; ST Elevation Myocardial Infarction
MeSH Terms: conditions — Sleep Apnea, Obstructive; ST Elevation Myocardial Infarction | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP treatment (Experimental): Continuous positive airway pressure (CPAP, AutoSet S9, ResMed, Sydney, Australia) plus standard care (according to current STEMI guidelines) for 3 months after pPCI
  Interventions: Device: Continuous positive airway pressure
- Control (No Intervention): Standard care (according to current STEMI guidelines) for 3 months after PPCI with no intervention for OSA

INTERVENTIONS:
Device: Continuous positive airway pressure — The optimal continuous positive airway pressure (CPAP, AutoSet S9, ResMed, Sydney, Australia) settings will be determined during 1-2 nights within 7 days after pPCI.
  Other Names: CPAP
  Arms: CPAP treatment

SUMMARY:
The aim of this randomized controlled trial to investigate the effects of CPAP treatment on myocardial salvage index and clinical outcomes at 3 months in patients with OSA and ST-Segment Elevation Myocardial Infarction (STEMI) after primary percutaneous coronary intervention (PPCI).

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years old
2. First-time STEMI
3. Successful PPCI (≥1 coronary artery) within 24h after symptom onset
4. Moderate to severe OSA (AHI≥15)
5. Written informed consent

Exclusion Criteria:

1. Prior myocardial infarction
2. Prior myocardial revascularization (PCI or CABG)
3. Cardiogenic shock (mean arterial pressure <60mmHg), severe heart failure (Killip≥3)
4. LM or multivessel disease indicated for CABG
5. History of stroke
6. Severe insomnia, chronic sleep deprivation, abnormal circadian rhythm (sleep <4h/night)
7. Severe COPD: FEV1/FVC <70% or FEV1 <50% predicted value (within 4 weeks)
8. Predominantly central sleep apnea (≥25% central events or central AHI ≥10/h)
9. Previous or current use of CPAP
10. Severe comorbidities: eg. malignancy (life expectancy <2 years)
11. Known or planned pregnancy
12. Known contraindication to CMR
13. Patients with contraindication to CPAP or who cannot tolerate it
14. Participation in other clinical trial in recent 3 months
15. Any condition that in the opinion of investigator that may jeopardize patient compliance, eg. significant memory, perceptual, or behavioral disorder, depression, severe alcohol consumption, or a history of noncompliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-03-26 (Estimated); Primary Completion 2019-03-24 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Myocardial salvage index | 3 months
  To investigate the effects of CPAP treatment on myocardial salvage index (MSI, assessed by cardiovascular magnetic resonance imaging, CMR) at 3 months in patients with OSA and ST-Segment Elevation Myocardial Infarction (STEMI) after primary percutaneous coronary intervention (PPCI)

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Ping NIE, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (2):
- China (2):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Undecided